CLINICAL TRIAL: NCT00392561
Title: Bangladesh Vitamin E and Selenium Trial
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Columbia University (Other); Dartmouth-Hitchcock Medical Center (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 15091A (R01-CA10743-1); AAAB2309 (Other: CUMC IRB)
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Non-melanoma Skin Cancer
MeSH Terms: interventions — Selenium; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Selenium
  Interventions: Dietary Supplement: Selenium
- 2 (Experimental): Vitamin E
  Interventions: Dietary Supplement: vitamin E
- 3 (Experimental): Vitamin E + Selenium
  Interventions: Dietary Supplement: Selenium; Dietary Supplement: vitamin E
- Arm 4 (No Intervention)

INTERVENTIONS:
Dietary Supplement: Selenium — 200 ug Selenium daily
  Arms: 1; 3
Dietary Supplement: vitamin E — 100 mg Vitamin E daily
  Arms: 2; 3

SUMMARY:
The purpose of this study is to evaluate whether selenium and/or vitamin E are effective in preventing non-melanoma skin cancers.

ELIGIBILITY:
Inclusion Criteria:

* Manifest arsenic skin lesions (melanosis, leucomelanosis, or keratosis)
* Aged 25 to 65 years
* Permanent resident of study area

Exclusion Criteria:

* Pregnancy
* Clinically too ill (enlarged spleen or liver)
* Presence of gangrene
* Cancer

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Skin Cancer | Incidence during the 6-year study period

SECONDARY OUTCOMES:
Mortality | Occurrence during the 6-year study period
Diabetes | Incidence within 6-year study period

CONTACTS AND LOCATIONS:
Overall Officials: Habibul Ahsan, MD, Principal Investigator — University of Chicago
Locations (2):
- Bangladesh (2):
  - Columbia University Arsenic Research Project, Dhaka
  - ICDDR,B, Dhaka

REFERENCES:
- [Derived] Jasmine F, Almazan A, Khamkevych Y, Argos M, Shahriar M, Islam T, Shea CR, Ahsan H, Kibriya MG. Gene-Environment Interaction: Small Deletions (DELs) and Transcriptomic Profiles in Non-Melanoma Skin Cancer (NMSC) and Potential Implications for Therapy. Cells. 2025 Jan 10;14(2):95. doi: 10.3390/cells14020095. PMID 39851523